CLINICAL TRIAL: NCT01142648
Title: The Effect of Sugammadex of EEG-derived Index Values
Brief Title: Sugammadex and Brain Waves
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Arvi Yli-Hankala/Professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R09041M; 2009-010916-14 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Anaesthesia
Keywords: Electroencephalogram; Electromyogram; Entropy Index; Bispectral Index; Reversal of neuromuscular blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 200 mg iv, single dose, bolus.
  Other Names: Bridion
Drug: Neostigmine and glycopyrrolate — Neostigmine 2.5 mg and glycopyrrolate 0,5 mg, iv, single dose, bolus, diluted in 2 ml volume with saline
  Other Names: Glycostigmin.

SUMMARY:
According to our experience, electroencephalogram-based indices of anaesthetic state show elevated numbers after administration of sugammadex (new reversal of neuromuscular blockade). This can be due to altered anaesthetic state, or some kind of artefact. In this study, the phenomenon is evaluated in detail.

DETAILED DESCRIPTION:
Rocuronium-induced neuromuscular blockade is antagonized with sugammadex or neostigmine. BIS, Entropy and the biosignal collected from the Entropy strip are collected on computer. The behaviour of these parameters before, during and after reversal on neuromuscular blockade will be analyzed in detail.

ELIGIBILITY:
Inclusion Criteria:

* females giving informed consent
* age range 18-65 years
* elective surgery: gynaecological
* general anaesthesia
* ASA classification 1 or 2

Exclusion Criteria:

* pregnancy
* body mass index > 30
* disease affecting CNS
* overuse of alcohol
* drug abuse
* unability to understand, read or use Finnish language

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The behaviour of depth of anaesthesia indexes (BIS,SE,RE) | 30 minutes

SECONDARY OUTCOMES:
The behaviour of electroencephalography | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, MD, Study Chair — Tampere University Hospital; Arvi Yli-Hankala, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland